CLINICAL TRIAL: NCT06990503
Title: An Open-label, Randomized, Multicenter Phase III Clinical Trial of SHR - A1811 Versus Investigator's Choice of Chemotherapy in the Treatment of Platinum-resistant Recurrent Epithelial Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer With HER2 Expression
Brief Title: SHR - A1811 Versus Chemotherapy for Platinum-resistant Recurrent Epithelial Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Prof., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-TJ-OVA1811R
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 Administration (Experimental): SHR-A1811 will be administered intravenously (IV) on Day 1 (D1) of each treatment cycle at a dose of 4.8 mg/kg. Treatment will be repeated every 3 weeks (one treatment cycle) , and will continue until the occurrence of any event meeting the protocol-defined criteria for treatment discontinuation.
  Interventions: Drug: SHR-A1811
- Chemotherapy Administration (Active Comparator): The investigator shall select one of the following treatment regimens (determined prior to randomization), and the treatment will be continued until the occurrence of any event meeting the protocol - defined criteria for treatment discontinuation.
  1. Liposomal doxorubicin Liposomal doxorubicin will be administered intravenously on Day 1 of each cycle at a dose of 40 mg/m², with one treatment cycle lasting 4 weeks.
  2. Paclitaxel Paclitaxel will be given intravenously on Days 1, 8, 15, and 22 of each cycle at a dose of 80 mg/m² per administration, and one treatment cycle is 4 weeks.
  3. Topotecan Topotecan will be administered intravenously on Days 1, 8, and 15 of each cycle at a daily dose of 4 mg/m², with a treatment - cycle duration of 4 weeks.
  4. Gemcitabine Gemcitabine will be infused intravenously on Days 1 and 8 of each cycle at a daily dose of 1000 mg/m², and each treatment cycle is 3 weeks.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: SHR-A1811 — Injection SHR - A1811 (hereinafter referred to as SHR - A1811) is an antibody - drug conjugate (ADC) targeting the HER2 protein, independently developed by Suzhou Shengdeya Biopharmaceutical Co., Ltd. (hereinafter referred to as the "sponsor"). It is composed of a recombinant humanized anti - HER2 IgG1 monoclonal antibody (SHR - 1805) conjugated with a small molecule component, SHR169106.
  Arms: SHR-A1811 Administration
Drug: Chemotherapy — The treatment regimens for the control group are as follows:
  Liposomal doxorubicin: Administered intravenously on Day 1 of each 4 - week treatment cycle at a dose of 40 mg/m².
  Paclitaxel: Given intravenously on Days 1, 8, 15, and 22 of each 4 - week treatment cycle at a dose of 80 mg/m² per administration.
  Topotecan: Intravenously infused on Days 1, 8, and 15 of each 4 - week treatment cycle at a daily dose of 4 mg/m².
  Gemcitabine: Infused intravenously on Days 1 and 8 of each 3 - week treatment cycle at a daily dose of 1000 mg/m².
  Arms: Chemotherapy Administration

SUMMARY:
This study is a randomized, open-label, active-controlled, multicenter phase III clinical trial.

It is planned to enroll 300 subjects with platinum-resistant recurrent epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer with HER2 expression. The randomization will be stratified according to the following factors: 1) HER2 immunohistochemistry (IHC) expression status (HER2 IHC 1+ versus HER2 IHC 2+/3+); 2) whether the subject has previously received vascular endothelial growth factor/vascular endothelial growth factor receptor (VEGF/VEGFR) inhibitors such as bevacizumab (yes versus no).

Subjects will be randomly assigned in a 1:1 ratio to receive either the experimental treatment group (SHR - A1811) or the control treatment group (chemotherapy chosen by the investigator, namely liposomal doxorubicin, paclitaxel, topotecan, or gemcitabine).

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in this trial and signs the informed consent form.
2. Female, aged 18 - 75 years old (including the boundary values, calculated from the date of signing the informed consent form).
3. Pathologically confirmed epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer by tissue or cytology.
4. Previously treated with a platinum - containing regimen and confirmed as platinum - resistant recurrence (platinum - resistant recurrence is defined as disease progression [PD] during platinum - containing therapy or within <183 days after the last dose of platinum - containing drugs). If the patient has only received 1 line of platinum - containing treatment, at least 4 cycles of platinum - containing drugs must be received. The determination of platinum - resistant recurrence must have clear documented radiological progression. After platinum resistance, at most 1 line of systemic anti - tumor treatment has been received, and the patient is suitable for single - agent chemotherapy in the next line of treatment.
5. Patients with known high expression of folate receptor α (FRα) must have received treatment with mirvetuximab soravtansine, unless the investigator judges that the patient is intolerant or unsuitable for mirvetuximab soravtansine treatment, or the treatment is not approved or unavailable locally, in which case they can be enrolled.
6. Disease progression during or after the last - line treatment, or toxicity that is intolerable (with clear evidence).
7. HER2 expression confirmed by the central laboratory: IHC 1+, 2+, or 3+; the patient needs to provide sufficient fresh or archived tumor tissue specimens for the sponsor - designated central laboratory to test the HER2 expression level (paraffin blocks, paraffin - embedded sections, or fresh tissue sections are all acceptable, and the scoring criteria for HER2 testing are determined by the central laboratory).
8. At least one measurable lesion that meets the RECIST v1.1 criteria (according to the RECIST v1.1 requirements, the long diameter of the measurable lesion on spiral computed tomography [CT] scan is ≥10 mm or the short diameter of the enlarged lymph node is ≥15 mm); lesions that have been locally treated can be selected as target lesions if there is clear evidence that they have significantly progressed compared with the post - treatment state.
9. ECOG PS score: 0 - 1 points.
10. Expected survival time ≥12 weeks.
11. Laboratory tests within 7 days before randomization confirm that the functions of important organs meet the following requirements (no blood components or cytokines can be used within 14 days before the tests):
12. Absolute neutrophil count ≥1.5×10⁹/L;
13. Platelet count ≥100×10⁹/L;
14. Hemoglobin ≥90 g/L;
15. Serum total bilirubin (TBIL) ≤1.5×the upper limit of normal (ULN);
16. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN;
17. Serum creatinine ≤1.25×ULN or creatinine clearance rate ≥50 mL/min (calculated according to the Cockcroft - Gault formula);
18. Activated partial thromboplastin time and international normalized ratio ≤1.5×ULN.
19. For female subjects of childbearing potential, the pregnancy test result during the screening period must be negative (if the investigator judges that a positive human chorionic gonadotropin [HCG] has no clinical significance and pregnancy is excluded, the subject can be included), and the subject must agree to use contraception and avoid donating eggs from the date of signing the informed consent form until 7 months after the last dose of IMP.

Exclusion Criteria:

1. Pathologically confirmed sarcoma histological subtypes, including hybrid tumors containing sarcomatous components.
2. Subjects with untreated or active central nervous system (CNS) tumor metastases. Subjects with a history of leptomeningeal metastasis or current leptomeningeal metastasis. Subjects whose CNS tumor metastases have undergone adequate local treatment (surgery or radiotherapy), do not require hormone therapy, have neurologically returned to baseline (except for residual signs or symptoms related to CNS treatment), and have been stable for ≥4 weeks can be enrolled.
3. Subjects who have previously received topoisomerase I inhibitors (including but not limited to irinotecan and topotecan), or ADC drugs containing topoisomerase I inhibitors, such as Enhertu (DS - 8201a), U3 - 1402, etc.
4. Subjects who have received systemic anti - tumor treatment within 4 weeks before the start of the study treatment. If the previous anti - tumor treatment was small - molecule targeted therapy, the interval between the end of treatment and the first study treatment should be no less than 5 half - lives of the drug or 7 days.
5. Subjects with symptomatic, poorly controlled, or moderate - to - severe pleural effusion, pericardial effusion, or ascites; subjects who have undergone effusion drainage (except diagnostic thoracentesis) can be enrolled if they have been stable for at least 2 weeks after drainage (local treatment within the serous cavity according to routine diagnosis and treatment is allowed before signing the informed consent form).
6. Subjects who have completed palliative radiotherapy within 7 days before the first dose.
7. Subjects with a history of other malignancies in the past or currently having other malignancies, except for cured basal cell carcinoma of the skin, cervical intraepithelial neoplasia, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, and other malignancies that have been adequately treated and cured for ≥3 years before randomization with evidence proving no recurrence or metastasis.
8. Subjects whose toxicity caused by previous anti - tumor treatment has not recovered to ≤Grade 1 according to the NCI - CTCAE v5.0 grading system (except for decreased lymphocyte count, alopecia, fatigue, and laboratory indicators mentioned in the inclusion criteria; some tolerable chronic Grade 2 toxicities can be excluded after consultation between the investigator and the sponsor).
9. Subjects with a history of interstitial pneumonia/interstitial lung disease or non - infectious pneumonia (such as radiation pneumonitis) that required steroid treatment; subjects with current or suspected interstitial pneumonia/interstitial lung disease, non - infectious pneumonia, or other active pneumonias; and subjects who experienced ≥Grade 3 interstitial pneumonia during previous treatment with immune checkpoint inhibitors.
10. Subjects with active pulmonary tuberculosis; subjects who have undergone adequate treatment before randomization and have stopped anti - tuberculosis treatment for ≥3 months can be enrolled.
11. Subjects with known pulmonary damage caused by concurrent pulmonary diseases, including but not limited to any potential pulmonary diseases (for example, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, etc. within 3 months before the first dose).
12. Subjects with autoimmune, connective tissue, or inflammatory diseases involving the lungs (such as rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.), or subjects who have previously undergone lobectomy or pneumonectomy.
13. Subjects with uncontrolled cardiac clinical symptoms or diseases, such as: (1) Heart failure of Grade 2 or above defined by the New York Heart Association (NYHA) criteria or left ventricular ejection fraction (LVEF) <50%; (2) Unstable angina; (3) Myocardial infarction within 1 year before randomization; (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) Fridericia - corrected QT interval (QTcF) >470 ms; (6) Hypertension that cannot be well controlled by drugs (subjects whose blood pressure is controlled at ≤160/100 mmHg with drugs can be enrolled).
14. Subjects who have experienced arterial or venous thrombotic events within 1 month before randomization, including but not limited to cerebrovascular accidents and deep vein thrombosis; subjects with intramuscular vein thrombosis or catheter - related thrombosis of the infusion port before randomization can be included if the investigator judges there is no risk.
15. Subjects who have experienced gastrointestinal perforation or fistula, urethral fistula, or abdominal abscess within 3 months before randomization; subjects who have undergone artificial fistulization or ureteral stent placement and are considered stable by the investigator after evaluation can be enrolled.
16. Subjects with intestinal obstruction or symptoms and signs of intestinal obstruction or those requiring parenteral nutrition within 3 months before the start of the study treatment. However, subjects who have undergone surgical treatment and the obstruction has been completely relieved can be screened; subjects who have previously undergone intestinal stent implantation and the stent has not been removed until the screening period.
17. Subjects who have experienced severe infections within 1 month before randomization, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc.; subjects with any active infections requiring intravenous systemic treatment, or subjects with unexplained fever >38.5°C during the screening period or before randomization.
18. Subjects with active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] test result during the screening period and hepatitis B virus - deoxyribonucleic acid [HBV - DNA] ≥500 IU/mL) or active hepatitis C (defined as positive hepatitis C virus [HCV] antibody test result during the screening period and positive HCV - ribonucleic acid [RNA]).
19. Subjects with a history of immunodeficiency, including positive human immunodeficiency virus (HIV) test results, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
20. Subjects who have undergone major surgery other than diagnostic or biopsy surgery within 28 days before the first dose; subjects who have undergone traumatic minor surgery (biopsy, laparoscopy, and drainage) within 7 days before the first dose; subjects with non - healing wounds (severe, non - healing, or dehisced wounds).
21. Subjects who are known to be allergic to any component of SHR - A1811; subjects with a history of severe allergic reactions to other monoclonal antibody fusion protein drugs.
22. Subjects with uncontrolled mental illness, known alcoholism, drug abuse, drug addiction, criminal detention, or other conditions that may affect the completion of the trial procedures.
23. Subjects with other serious diseases, including but not limited to acute myocardial infarction within the past 3 months, acute cerebral infarction within the past 3 months, decompensated cirrhosis, etc.
24. Other conditions that, in the opinion of the investigator, may increase the risk of participating in the trial, interfere with the trial results, or make the subject unsuitable for this trial.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian cancer patients
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 5 Years after treatment.
  Progression - Free Survival (PFS) as assessed by the Independent Radiological Review Committee (IRC) based on the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). It is defined as the time from the randomization date of the subject to the first date of documented radiological tumor progression or the date of death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 Years after treatment.
  Defined as the time from the randomization date to death due to any cause in subjects.
Objective Response Rate (ORR): | 5 Years after treatment.
  Defined as the proportion of subjects who achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) as assessed by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). For responses categorized as CR or PR, confirmation is required through a subsequent evaluation performed no less than 4 weeks (≥28 days) after the initial assessment.
Duration of Response (DoR) | 5 Years after treatment.
  Defined as the time from the first date a subject is assessed as having a confirmed Complete Response (CR) or Partial Response (PR) to the first date of either Progressive Disease (PD) or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 5 Years after treatment.
  Defined as the proportion of subjects with a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as assessed by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Response Rate (RR) | 5 Years after treatment.
  Defined as the proportion of subjects with an overall response assessed as either a response according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or a response according to the Gynecologic Cancer InterGroup (GCIG) CA - 125 criteria.
CA - 125 Response Rate (CA - 125 RR) | 5 Years after treatment.
  Defined as the proportion of subjects with a response evaluated according to the Gynecologic Cancer InterGroup (GCIG) CA - 125 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Gao for primary data.